CLINICAL TRIAL: NCT05198245
Title: Retrospective Cohort Study of Pregnancy Outcomes in Women Exposed to Rimegepant During Pregnancy
Brief Title: Study of Pregnancy Outcomes in Women Exposed to Rimegepant During Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: RTI Health Solutions (Other); Optum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV3000-403; C4951006 (Other: Alias Study Number)
Record Dates: First submitted 2021-12-15; First posted 2022-01-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Migraine Disorder; Migraine Prevention; Prevention of Migraine; Pregnant; Pregnancy; Infant
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnancies in women with migraine and exposure to rimegepant
  Interventions: Drug: Rimegepant
- Pregnancies in women with migraine exposed to other medications: Pregnancies in women with migraine exposed to other medications indicated for the treatment of migraine
  Interventions: Drug: Various
- Pregnancies in women without migraine
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75mg
  Groups: Pregnancies in women with migraine and exposure to rimegepant
Drug: Various — Various
  Groups: Pregnancies in women with migraine exposed to other medications
Other: No intervention — No intervention
  Groups: Pregnancies in women without migraine

SUMMARY:
The purpose of the study is to evaluate the risk of pregnancy and infant outcomes among women with migraine exposed to rimegepant during pregnancy and in two rimegepant unexposed comparator groups.

ELIGIBILITY:
Inclusion Criteria (All Pregnancies):

All pregnant women aged 16 to 49 years, inclusive, at the estimated LMP within the study observation period are eligible to enter in the study.

Exclusion Criteria (All Pregnancies):

* Has insufficient information to estimate LMP
* Has at least 1 pharmacy dispensing for ditans (i.e., lasmiditan) within a 5-half-life time window before the estimated LMP through whichever is first: end of pregnancy or end of the study period
* Has at least 1 pharmacy dispensing for a CGRP receptor antagonist other than rimegepant (i.e., ubrogepant, atogepant, and zavegepant) within a 5-half-life time window before the estimated LMP through whichever is first: end of pregnancy or end of the study period
* Has at least 1 pharmacy dispensing for CGRP monoclonal antibodies (i.e., erenumab, fremanezumab, eptinezumab, and galcanezumab) within a 5-half-life time window before the estimated LMP through whichever is first: end of pregnancy or end of the study period

Additional Eligibility Criteria (Rimegepant-Exposed Group):

* Have a migraine diagnosis any time before the estimated LMP and through whichever is first: end of pregnancy or end of the study period
* Have at least 1 pharmacy dispensing for rimegepant within the 30-day time window before the estimated LMP and through whichever is first: end of pregnancy or end of the study period
* Have a recorded outcome of pregnancy within the study period
* Had continuous enrollment in a health care plan with medical and pharmacy benefits during the 6-month period before the estimated LMP through a postpartum period of 42 days

Additional Inclusion Criteria (Primary Comparator Group):

* Have a migraine diagnosis any time before the estimated LMP and through whichever is first: end of pregnancy or end of the study period
* Have at least 1 pharmacy dispensing for a medication indicated for the treatment of migraine within the 30-day time window before the estimated LMP and ending with whichever is first: end of pregnancy or end of the study period.
* Have a recorded outcome of pregnancy within the study period
* Had continuous enrollment in a health care plan with medical and pharmacy benefits during the 6-month period before the estimated LMP through a postpartum period of 42 days

Additional Exclusion Criteria (Primary Comparator Group):

• Have at least 1 pharmacy dispensing for rimegepant within the 30-day time window before the estimated LMP and through whichever is first: end of pregnancy or end of the study period

Additional Inclusion Criteria (Secondary Comparator Group):

* Have no migraine diagnosis any time before the estimated LMP through whichever is first: end of pregnancy or end of the study period
* Have a recorded outcome of pregnancy within the study period
* Had continuous enrollment in a health care plan with medical and pharmacy benefits during the 6-month period before the estimated LMP through a postpartum period of 42 days

Additional Exclusion Criteria (Secondary Comparator Group):

• Have at least 1 pharmacy dispensing for rimegepant within the 30-day time window before the estimated LMP through whichever is first: end of pregnancy or end of the study period

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will consist of pregnant women (any age) as well as the infants (male and female) born to enrolled participants through age 1 year
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformations, spontaneous abortions, fetal deaths/stillbirths, small for gestational age births | Annually beginning April 2022

SECONDARY OUTCOMES:
Elective terminations | Annually beginning April 2022
Preterm births | Annually beginning April 2022
Pre-eclampsia/eclampsia | Annually beginning April 2022

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-403